CLINICAL TRIAL: NCT05981599
Title: Epidemiological, Clinical and Biological Caracteristics of Patients Presenting With Invasive Meningococcal Disease in the West of France
Brief Title: Epidemiological, Clinical and Biological Caracteristics of Patients Presenting With Invasive Meningococcal Disease
Acronym: CARACIIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CARACIIM
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Meningococcal Infections
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention. Only retrieving clinical, biological and epidemiological data from patient files

SUMMARY:
An unusual increase in cases of invasive meningococcal infection between late 2022 and early 2023. These cases sometimes had atypical presentations (large numbers of bacteremias without meningitis). The distribution of serogroups was also unusual in our center (large number of serotype Y meningococcal IMD).

This development comes after three years marked by the Corona-Virus-Disease-19 pandemic, which led to a profound change in the behaviors involved in the transmission of infectious diseases. Barrier measures have considerably reduced the population's exposure to meningococcus, and may have encouraged a reduction in mucosal immunity to this pathogen. The end of 2022 was also marked by intense viral circulation (syncitial respiratory virus-influenza-COVID), which may have favored invasive forms.

DETAILED DESCRIPTION:
Invasive meningococcal disease (IMD) accounts for a small number of cases (500-600 cases/year) in mainland France. Despite advances in its management, the disease is still associated with a 10-20% mortality rate and impaired quality of life in 50% of surviving patients.

An unusual increase in cases of invasive meningococcal infection during the winter of 2022. These cases often had atypical presentations (large number of bacteremias without meningitis, digestive picture in the foreground). The distribution of serogroups was also unusual at our center (large number of serotype Y meningococcal IMD). These data appear to be confirmed by Santé Publique France's national data for 2022, with no warning of the spread of a hyper-virulent clone.

This development comes after three years marked by the SARS-CoV2 pandemic, which led to a profound change in the behaviors involved in the transmission of infectious diseases .

Barrier measures have considerably reduced the population's exposure to meningococcus, and may have led to a reduction in mucosal immunity to this pathogen. This is particularly true of teenagers and young adults, for whom contact has fallen sharply due to the closure of schools and universities. It would be interesting to see whether this population is more affected this year than in previous years.

The end of 2022 was also marked by intense viral circulation (SRV-Flu-Covid), which could have favored invasive forms. Evidence of a significant number of viral co-infections could support this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Invasive Meningococcal infection (defined by the isolation of Neisseria meningitis in a normaly steril site (CSL, blood, articulation, ..) by PCR or culture.

No exclusion Criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient from the West part of France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient presenting with Invasive Meningococcal infection and its serogroup | Two period of 18month, one when facial mask were recommanded, and one after
  - Evolution of the Number of case according to time and the evolution of serogroup There will be two study period. The number of Invasive Meningococcal infection and their serogroup will be counted in each period.

CONTACTS AND LOCATIONS:
Overall Officials: France CAZENAVE ROBLOT, PhD, Study Director — SPILF
Locations (1):
- Poitiers University, Poitiers, Vienne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Actuality report — https://www.santepubliquefrance.fr/content/download/504135/3759948?version=2 — French Report on the epidemic situation of meningococcal disease in december 2022
- Available data/document: Clinical Study Report — https://doi.org/10.1371/journal.pone.0281544